CLINICAL TRIAL: NCT01077960
Title: Phase III, Multi-Center, Open, 12-Week, Follow-up Safety and Efficacy Study of Serostim® in Subjects With Human Immunodeficiency Virus-Associated Adipose Redistribution Syndrome (HARS)
Brief Title: Safety and Efficacy Study of Serostim® Human Immunodeficiency Virus-Associated Adipose Redistribution Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25373 (NCT01077960)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Results first posted 2010-06-23 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Human Immunodeficiency Virus-Associated Adipose Redistribution Syndrome
Keywords: Serostim; HARS
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Serostim (Experimental): Serostim® 4 mg daily given for 12 weeks (following a prior 36-week treatment [Serono Study 24380] with Serostim® 4 mg daily given for 12 weeks, followed by 24-weeks of either Serostim® 2 mg every other day or Placebo every other day)
  Interventions: Biological: Serostim

INTERVENTIONS:
Biological: Serostim — Serostim® 4 mg daily given for 12 weeks (following a prior 36-week treatment [Serono Study 24380] with Serostim® 4 mg daily given for 12 weeks, followed by 24-weeks of either Serostim® 2 mg every other day or Placebo every other day)
  Other Names: mammalian cell-derived recombinant human growth hormone; r hGH

SUMMARY:
In Serono Study 24380, the antecedent protocol to Study 25373, patients were randomly assigned in a 3.0-to-1.0 ratio to Groups A and B. All patients in Group A received recombinant human growth hormone (Serostim®) 4 mg daily (the "induction" phase) for the first 12 weeks, and then were re-randomized to receive either placebo or Serostim 2 mg on alternate days (roughly equivalent to 1 mg daily) during Weeks 12-36 (the "maintenance" phase). All patients in Group B initially received placebo from baseline to Week 24, and then received Serostim® 4 mg daily from Weeks 24 to 36 (Grunfeld, 2007).

In the follow-up Study 25373, any subject who was enrolled in Serono Study 24380 and was assigned to Group A, who fully completed all study visits without a major protocol violation, was eligible to enroll to receive re-treatment with Serostim at a dose of 4 mg daily for 12 weeks. During study 25373, safety was monitored by recording of adverse events and measurement of urinalysis and laboratory blood tests to assess fasting glucose, fasting insulin, and routine biochemistry and hematology parameters. At Week 12 or at the time of study termination, subjects underwent re-assessment of body composition via anthropometry measurements and dual photon absorptiometry (DXA) scanning. In addition, at study termination, measurements of insulin-like growth factor I (IGF-I), insulin-like growth binding protein 3 (IGFBP-3), fasting lipid profile, and oral glucose tolerance testing were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Must meet all inclusion/exclusion criteria for Serono Study 25373, have participated in Serono Study 24380, must have been assigned to Group A, must have completed all treatments and procedures (including baseline, Week 12 and Week 36 Computerized Tomography (CT) and Dual-Energy X-ray Absorptiometry (DXA) Scans) and had no major protocol violation.
* Must be taking antiretroviral medications that are approved or are available under a Treatment Investigational New Drug (IND). Subjects must also agree not to discontinue or to change their regimen for the duration of the study except as judged medically necessary.
* Must be willing and able to comply with the protocol for the duration of the study.
* Must have voluntarily provided written informed consent and a subject authorization under Health Insurance Portability and Accountability Act of 1996 (HIPAA), prior to any study-related procedure that is not part of normal medical care, and with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.
* If female, subjects must either:

  * Be post menopausal (=/>1 year) or surgically sterilized (i.e., have undergone tubal ligation or hysterectomy), or
  * Use a contraceptive method for the duration of the study such as: hormonal contraceptive,intra uterine device,diaphragm with spermicide, or condom with spermicide, and
  * Must be neither pregnant nor breast feeding.
  * Confirmation that female subjects of childbearing potential are not pregnant must be established by a negative pregnancy test prior to initiating first treatment.

A pregnancy test is not required if the subject is post menopausal or surgically sterilized.

Exclusion Criteria:

* Have any condition, which interferes with informed consent or protocol compliance including, but not limited to, active substance abuse and/or dementia.
* Have any active malignancy, except localized cutaneous Kaposi's sarcoma (fewer than 10 lesions, none of which are larger than 2 cm, and not on active therapy).
* Have active central nervous system (CNS) process associated with neurological findings.
* Have acute illness treated in an intensive care unit, e.g., due to complications following open heart or abdominal surgery, multiple accidental trauma, or acute respiratory failure.
* Have any medical condition in view of which the study doctor and/or Serono Medical/Therapeutic Director feels that it would be in the best interest of the subject not to participate in the follow-up study.
* Are unable to comply with the Concomitant Therapy restrictions as outlined in Section 5.5 and listed as follows:

  * Therapy for obesity including therapy with anorexigenic or fat reducing drugs.
  * Anti-diabetic or insulin sensitizing medications.
  * Systemic glucocorticoids.
  * Systemic chemotherapy, interferon or radiation therapy treatment.
  * Androgenic agents including, but not limited to, testosterone, nandrolone (Deca-durabolin), oxandrolone (Oxandrin), oxymetholone (Anadrol), dehydroepiandrosterone (DHEA), etc. (Testosterone replacement therapy for hypogonadism is the exception to this exclusion and will be allowed if started >30 days prior to Study Day 1 of Serono Study 24380).
  * Progestational agents, unless used for oral contraception or post-menopausal hormone replacement therapy.
  * Appetite stimulants such as dronabinol (Marinol), megestrol acetate (Megace), or cyproheptadine (Periactin).
  * Investigational agents, unless approved in advance by Serono's Medical Director. Specifically, experimental antiretroviral agents are disallowed, unless available under a treatment IND or expanded access program (30 days).
  * Liposuction or other elective plastic surgery.
  * Acquired Immune Deficiency Syndrome (AIDS) wasting therapy with growth hormone and/or prior treatment with growth hormone or a growth hormone releasing factor (for 12 months prior to the screening visit).
* Are participating in any other clinical studies (except Serono Study 24380). Observation studies are allowed, but prior written permission by Serono Medical/Therapeutic Director must be granted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-02; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (25):
  - University of Alabama/Birmingham, Birmingham, Alabama
  - Care Clinic, Los Angeles, California
  - Private Practice, Palm Beach, California
  - UCSD - AVRC (AntiViralResearchCenter), San Diego, California
  - Kaiser Permanente, San Francisco, California
  - Harbor-UCLA Medical Center, Torrence, California
  - AIDS Alliance, West Hollywood, California
  - Circle Medical LLC, Norwalk, Connecticut
  - Private Practice, Washington D.C., District of Columbia
  - Private Practice, Fort Lauderdale, Florida
  - Care Resources, Miami, Florida
  - Private Practice, Miami, Florida
  - Private Practice, North Miami Beach, Florida
  - Infectious Disease Associates, Sarasota, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Community Research Initiative of New England, Boston, Massachusetts
  - Tufts University School of Medicine, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - St. Luke's Roosevelt Hospital, New York, New York
  - St. Vincents Catholic Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Central Texas Clinical Research, Austin, Texas
  - IPD Research, Annandale, Virginia
  - Private Practice, Spokane, Washington
- St Paul Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Grunfeld C, Thompson M, Brown SJ, Richmond G, Lee D, Muurahainen N, Kotler DP; Study 24380 Investigators Group. Recombinant human growth hormone to treat HIV-associated adipose redistribution syndrome: 12 week induction and 24-week maintenance therapy. J Acquir Immune Defic Syndr. 2007 Jul 1;45(3):286-97. doi: 10.1097/QAI.0b013e3180691145. PMID 17592343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date: 03 Feb 2005 (date of first subject, first dose) Study Completion Date 04 Jan 2006 (date of last subject, last visit) 26 study centers in the United States and British Columbia participated in this study, with each center enrolling at least one subject into the study.
Pre-assignment Details: Any subject who was enrolled in Serono Study 24380, assigned to Group A, and fully completed all study visits without major protocol violations was to be allowed to enroll in Study 25373
Period: Overall Study
Arm/Group | Serostim
Started | 126 (130 subjects consented to participate, 129 enrolled in the study, and 126 received study drug)
Completed | 110 (Modified Intent To Treat (ITT) Population)
Not Completed | 16
Not completed — Adverse Event | 6
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 5
Not completed — Subject decision | 1
Not completed — Reason unspecified | 1

BASELINE CHARACTERISTICS:
Arm/Group | Serostim
Number analyzed (Participants) | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 126
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 113
Region of Enrollment [Number; unit: participants]
  United States | 125
  Canada | 1
Insulin-like Growth Factor I [Mean (Standard Deviation); unit: ng/mL] — n=112
  ng/mL | 242.6 (132.8)
Oral Glucose Tolerance Testing - 120 Minute Glucose [Mean (Standard Deviation); unit: mg/dL] — n=105
  mg/dL | 102.3 (35.7)
Oral Glucose Tolerance Testing - Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] — n=124
  mg/dL | 94.5 (14.7)
Oral Glucose Tolerance Testing - Fasting Insulin [Mean (Standard Deviation); unit: mcIU/mL] — n=111
  mcIU/mL | 11.4 (13.6)
Trunk Fat [Mean (Standard Deviation); unit: kg] — n=106
  kg | 10.4 (4.9)
Waist Circumference [Mean (Standard Deviation); unit: cm] — N=116
  cm | 97.3 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Trunk Fat as Assessed by Dual-Energy X-Ray Absorptiometry (DXA) Scan
Time Frame: baseline to 12 weeks
Population: The analysis population reported here comprised the subjects who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Serostim
Number analyzed (Participants) | 106
kg | -1.7 (1.4)
Statistical Analysis 1: Comparison: Serostim; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Change From Baseline to Week 12 in Waist Circumference
Description: Measured by anthropometry
Time Frame: baseline to 12 weeks
Population: The analysis population reported here comprised the subjects who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Serostim
Number analyzed (Participants) | 116
cm | -1.5 (3.0)
Statistical Analysis 1: Comparison: Serostim; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Change From Baseline to Week 12 in Insulin-like Growth Factor I
Description: Circulating levels of IGF-I
Time Frame: baseline to 12 weeks
Population: The analysis population reported here comprised the subjects who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Serostim
Number analyzed (Participants) | 112
ng/mL | 135.7 (210.7)
Statistical Analysis 1: Comparison: Serostim; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Oral Glucose Tolerance Testing - Change From Baseline to Week 12 in Fasting Insulin
Description: Oral glucose tolerance testing
Time Frame: baseline to 12 weeks
Population: The analysis population reported here comprised the subjects who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: mcIU/mL
Arm/Group | Serostim
Number analyzed (Participants) | 111
mcIU/mL | 10.8 (22.3)
Statistical Analysis 1: Comparison: Serostim; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Oral Glucose Tolerance Testing - Change From Baseline to Week 12 in 120 Minute Glucose
Description: Oral glucose testing
Time Frame: baseline to 12 weeks
Population: The analysis population reported here comprised the subjects who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Serostim
Number analyzed (Participants) | 105
mg/dL | 11.7 (43.7)
Statistical Analysis 1: Comparison: Serostim; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

6. Secondary Outcome: Oral Glucose Tolerance Testing - Change From Baseline to Week 12 in Fasting Glucose
Description: Oral glucose testing
Time Frame: baseline to 12 weeks
Population: The analysis population reported here comprised the subjects who received at least one dose of study drug
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Serostim
Number analyzed (Participants) | 124
mg/dL | 4.5 (20.4)
Statistical Analysis 1: Comparison: Serostim; Test type: Superiority or Other; p = 0.015, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were to be reported and collected on an ongoing basis from the day of written informed consent (baseline) until 4 weeks after the last investigational product administration.
Description: Adverse events occurring during study treatment are reported
Arm/Group | Serostim
Serious Adverse Events (participants affected / at risk) | 2/126
Other Adverse Events (participants affected / at risk) | 89/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Serostim (N=126)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Serostim (N=126)
Oedema peripheral (General disorders) | 31 (47)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (30)
Hypoaesthesia (Nervous system disorders) | 9 (9)
Blood glucose increased (Investigations) | 8 (8)
Joint swelling (Musculoskeletal and connective tissue disorders) | 8 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (7)
Insomnia (Psychiatric disorders) | 7 (7)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 7 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other